CLINICAL TRIAL: NCT04630912
Title: Acceptance and Commitment Therapy (ACT) for People With Dementia Experiencing Psychological Distress: a Hermeneutic Single Case Efficacy Design (HSCED) Series
Brief Title: ACT for People With Dementia Experiencing Psychological Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Nottinghamshire Healthcare NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20064
Record Dates: First submitted 2020-11-02; First posted 2020-11-16 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Acceptance and Commitment Therapy; Dementia
Keywords: Dementia; Psychological distress; Psychological therapy; ACT; Acceptability; HSCED
MeSH Terms: conditions — Dementia | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Hermeneutic single case efficacy design (HSCED) series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acceptance and Commitment Therapy (Experimental): 12 weekly, 90 minute ACT sessions with person with dementia (with a review at week 6)
  Interventions: Other: Acceptance and Commitment Therapy

INTERVENTIONS:
Other: Acceptance and Commitment Therapy — There is no specific protocol for ACT with dementia, therefore a published ACT protocol, 'Better Living with Illness' (Brassington et al., 2016), will be used flexibly to guide the intervention.

SUMMARY:
Introduction: People with dementia have a high prevalence of psychological distress but are under-served with evidence-based psychological interventions. To promote choice and improve clinical outcomes, there is a necessity to test different psychological intervention options for this population. Purpose: To investigate the effectiveness and acceptability of Acceptance and Commitment Therapy (ACT) for people with dementia, considering carer-supported, remote delivery and necessary therapy adaptations. Methods: A hermeneutic single case efficacy design (HSCED) series was used to analyse therapy process and change for three clients with dementia and psychological distress. Quantitative and qualitative data was collated ('rich case records') and analysed by three independent psychotherapy experts ('judges') who determined the outcome for each client. Results: Over the course of therapy, it was concluded that one client with dementia made positive changes, specifically reliable reductions in psychological distress, which were largely attributable to Acceptance and Commitment Therapy (ACT). Two clients remained unchanged. Discussion/Conclusion: Where change was achieved, the ACT-specific processes of values, committed action and acceptance, in combination with non-specific therapy factors including a strong client-carer relationship, existing client interests and individualised therapy adaptations, were facilitative of change. Hence, ACT may be feasible and effective by helping carers to better meet the needs of their loved ones with dementia. Future research to optimise ACT delivery in this population may be beneficial. Furthermore, the assessment of carer factors (e.g., their psychological flexibility, the client-carer relationship) may strengthen the evidence-base for systemic ACT-use.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for people with dementia

Participants were included in the study if they had:

* A clinical diagnosis of dementia (any type)
* A clinically significant level of psychological distress (a score of ≥8 on the GAD-7 and ≥10 on the PHQ-9).
* Ability to give informed consent

Inclusion criteria for caregiver of person with dementia

Participants were included in the study if they:

* Cared for someone with a clinical diagnosis of dementia (any type)
* Were paid or unpaid and regularly supported them with activities of daily living
* Aged 18+ (no maximum age limit)
* Able to give informed consent

Exclusion Criteria:

Exclusion criteria for people with dementia

Participants were excluded if they:

* Were already receiving psychotherapy
* Had insufficient English or language abilities to engage in therapy
* Were unable to consent to and/or engage in therapy

Exclusion criteria for caregiver of person with dementia

Participants were excluded if they:

* Had insufficient English or language abilities to support the person with dementia or engage in study/Change Interviews
* Were unable to consent to and/or engage in study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Change in anxiety | Through study completion, up to 24 weeks
  Generalised anxiety disorder questionnaire (GAD-7), scored 0-21, where higher scores indicate a greater severity of anxiety.
Change in depression | Through study completion, up to 24 weeks
  Patient health questionnaire (PHQ-9), scored 0-27, where higher scores indicate a greater severity of depression.

SECONDARY OUTCOMES:
Change in psychological flexibility | Through study completion, up to 24 weeks
  Comprehensive assessment of Acceptance & Commitment Therapy (CompACT-SF), scored 0-48, where higher scores indicate increased psychological flexibility.
Change in wellbeing | Through study completion, up to 24 weeks
  Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWS), scored 7-35, where higher scores indicate higher mental wellbeing.
Change in client problems | Through study completion, up to 24 weeks
  Personal questionnaire (PQ), where higher scores indicate greater severity of problems.
Change in therapeutic alliance | Through study completion, up to 12 weeks
  Session rating scale (SRS), does not involve numerical values but asks clients to mark on a line nearest to the description that best fits their experience (marks further towards the right indicate better therapeutic alliance).

CONTACTS AND LOCATIONS:
Overall Officials: Danielle De Boos, Dr, Study Director — University of Nottingham
Locations (1):
- Community Mental Health Team for Older People, Newark, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The study data was written up as part of the student Doctoral Thesis and will be submitted in partial fulfilment of the requirements for the Trent Doctorate in Clinical Psychology (DClinPsy) in February 2022.
  Participants chose a pseudonym for themselves to be used in publications (e.g. electronic documents, written notes and transcripts) to prevent identification and references to personal information (e.g. other people's names, locations) were altered.
Supporting Information: CSR
Time Frame: July 2022